CLINICAL TRIAL: NCT07033988
Title: Insights Into Cerebral Clot Biomarkers and Inflammatory Pathways
Brief Title: Study of Inflammatory Cells in the Blood and Cerebral Thrombus of Patients Affected by Cerebral Ischemia
Acronym: ClotBioInsight
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: University of Zurich (Other); University of Manchester (Other); German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Bacigaluppi Marco, Principal Investigator, IRCCS San Raffaele
Other Study IDs: CET 96-2025
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Stroke Acute
Keywords: stroke; thrombectomy; clot; inflammation; biomarker; pathphysiology
MeSH Terms: conditions — Stroke; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cerebral thrombus and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke_Patients: This cohort includes adult patients diagnosed with acute ischemic stroke due to large vessel occlusion (LVO); subgroups within the cohort may include patients with different etiologies based on standard diagnostic classifications and stratification may be performed by response to thrombolysis, histological thrombus composition, or systemic biomarkers.

SUMMARY:
This is an observational, prospective and retrospective, single-center study of thrombotic material and blood samples obtained from patients undergoing mechanical endovascular thrombectomy for ischemic stroke caused by large vessel occlusion or stenosis.

The overarching aim of this study is to advance the understanding of the pathogenesis of cerebral ischemia and to support the development of novel therapeutic strategies for cerebrovascular disease. Specifically, the research seeks to elucidate the pathophysiological mechanisms involved in thrombus formation and stabilization that lead to ischemic events, identify thrombus compositions associated with distinct stroke etiologies, and determine features predictive of resistance to current intravenous thrombolytic therapies. In addition, the study aims to discover novel therapeutic targets and to identify circulating blood biomarkers indicative of an elevated risk of thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Presentation to the emergency department with symptoms and/or signs suggestive of:
* An acute cerebrovascular event
* Stroke mimics
* Stroke-related risk factors (e.g., atrial fibrillation, endocarditis, significant internal carotid stenosis, neoplasms, systemic infections)
* Undergoing one of the following treatments:
* Mechanical thrombectomy
* Intravenous thrombolysis
* Standard medical therapy
* Provision of informed consent, either:
* Directly from the conscious patient
* Via appropriate procedures for unconscious patients

Exclusion Criteria:

* Pregnancy or breastfeeding
* Presence of a known autoimmune disease that could interfere with the interpretation of biomarker analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study focuses on adult patients experiencing ischemic stroke presenting at the emergency department/ neurology department of the Hospital of inclusion due to a large vessel occlusion and/or stenosis, undergoing standard diagnostic and therapeutic procedures involving mechanical thrombectomy, thrombolysis or standard medical care.
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Quantification of leukocyte Infiltration in Thrombus | 01.07.2025 up to 06.05.2030
  Leukocyte will be quantified in thrombus sections using immunohistochemistry or immunofluorescence staining for neutrophil markers such as CD45, Cd11b, etc..
Assess the number of neutrophil extracellular traps (NETS) | from 6/2025 to 5/2030
  NETs will be quantified in thrombus tissue sections using immunofluorescence staining for citrullinated histone H3 and myeloperoxidase (MPO).

SECONDARY OUTCOMES:
Quantitative Analysis of Red Blood Cells, Fibrin, von Willebrand Factor, and Platelets in Thrombus. | 01.08.2025 - 01-05-2030
  Histological components of the thrombus-including red blood cells (RBCs), fibrin, von Willebrand factor (vWF), and platelets-will be evaluated using immunohistochemistry and immunofluorescence staining. Quantification will be expressed as percentage area fraction (% of total thrombus area) occupied by each component, as assessed by digital image analysis of stained slides.
Quantification of Plasma Cytokine Levels in Ischemic Stroke Patients | 01.08.2025 - 01.05.2030
  Plasma cytokines will be measured using multiplex immunoassays or ELISA-based methods from peripheral blood samples collected during the acute and subacute phases of ischemic stroke. Concentrations (pg/mL) of cytokines will be quantified and reported as continuous variables to assess systemic inflammatory responses.

OTHER OUTCOMES:
Characterization of Circulating and Tissue-Derived Cell Populations | 01.08.2025 - 01.05.2030
  Cellular profiles will be analyzed from peripheral and tissue-derived samples using advanced molecular and analytical techniques. Data will include single- sell level measurements to explore cellular heterogeneity and potential pathological signatures, summarized by relative abundance and classification of major cell populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No